CLINICAL TRIAL: NCT04407884
Title: Long Term Use of a High Energy Pulsed Heating Device in the Management of Chronic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soovu Labs Inc. (Industry)
Responsible Party: Principal Investigator, charles chabal, Chief Science officer, Soovu Labs Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soovu 001-20
Record Dates: First submitted 2020-05-17; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Pain; Pain, Chronic; Pain, Back
Keywords: heat; analgesia; chronic pain; thermal analgesia; low back pain
MeSH Terms: conditions — Pain; Chronic Pain; Back Pain; Agnosia; Low Back Pain

STUDY DESIGN:
Intervention Model Description: Single group with longitudinal follow-up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study arm (Experimental): Subjects will receive an active study device.
  Interventions: Device: Soovu Labs Inc. Pain Relief System

INTERVENTIONS:
Device: Soovu Labs Inc. Pain Relief System — Longnitual follow-up

SUMMARY:
The purpose of this study is to evaluate the Soovu Labs pain Relief System in a group of users that represent people most likely to purchase and use the units. This study is called an In Home Users Trial (IHUT). The device is called Soovu and was determined by the FDA to be Class II 510(k) except (C190061 November 2019). Relevant endpoints include ease of use, pain relief, quality of life, and long-term effectiveness.

DETAILED DESCRIPTION:
Soovu device description:

From the FDA document (C190061) "The system is indicated to provide topical heating for the purpose of elevating tissue temperature for the temporary relief of minor muscle and joint pain and stiffness; the temporary relief of joint pain associated with arthritis; the temporary relief of muscle spasms, minor sprains and strains, and minor muscular back pain; the temporary relief of menstrual discomfort; the relaxation of muscles; and the temporary increase of local circulation where applied." The devices are constructed following documented ANSI/AAMI ES60601-1, ANSI/AAMI HA60601-1-11, IEC 60601-1-2, IEC 60529, ISO 10993-5, and 10993-10 safety standards.

The device consists of two separate heating units pods that are attached to the body via a ring coated with medical grade adhesive. The units are easily removed from the body. The units are controlled by a phone app that the user downloads to his or her phone and pairs with the units via Bluetooth. The app contains instructional material on how to use the device and general information related to pain management. The user may start and end heat cycles via the app, may adjust the temperature of the unit, and select from one of three heating profiles. The maximum temperature of the unit is 113° F well within accepted safety limits. The three heating algorithms are:

1. Waves of heat up 113F that occur about 2 times per minute for up to 30 minutes
2. Waves of heat up 113F that occur about 4 times per minute for up to 30 minutes
3. Waves of heat up 113 F that occur about 2-3 times per minute for up to 30 minutes. These waves of heat are synchronized with instructions in the app that guide users through relaxed breathing exercises sometimes called box breathing. This option lasts up to 30 minutes.

The user can freely select any of the options, can end the session before the 30 minute time out, and can reduce the maximum temperature of the heat wave from 113° F all via the app.

Objective(s) To assess the consumer experience of Soovu Labs wearable thermal pulsed-heat device with Blue-tooth connected app among patients with recurring lower back. Assessment will include a) whether the device is perceived to work in managing their pain, b) if the device is comfortable to wear and use, c) if the app is easy to use, and d) if patients would purchase the product and replacement adhesive.

Design Single arm. home-use study

Treatment Participants will be provided with a Soovu Labs device. Back pain sufferers will apply the product to their pain site as needed following label instructions during an approximate 60 day usage period. Participants will download the app to their personal mobile phone.

Number of Patients A total of 40 participants will be recruited for the study.

Rationale Pain is an unpleasant sensory and emotional experience that is associated with actual or potential tissue damage or is described associated with such damage. It causes significant disability and dramatically decreases the patients' quality of life especially if it lasts for a long time and becomes chronic. Many key opinion leaders and experts in orthopedics and rheumatology accept that the pain is considered chronic if it lasts more than six months. Chronic neck, back, and shoulder pain are among the most common and disabling conditions accompanying different musculoskeletal disorders. As many other chronic painful conditions, they are very disabling and lead to considerable stress on healthcare systems. Several treatment modalities and their combinations have been proposed with different success rates, including exercises, physical therapy, oral medication, injections and even surgery. However, many products have low satisfaction rates given poor design, poor aesthetics, and limited effectiveness.

The present study suggests a new therapeutic option (pulsed heat) for patients with recurring lower back or cervical pain. The new wearable device delivers pulsed heat that automatically raises and lowers the heat intensity over wear time may provide a better patient experience. This study will assess opinions of likely users about the device.

Study Procedures The IHUT study will be run by Soovu Labs Inc. Seattle, WA.

Subjects may be recruited via an internal database of those who have participated in previous studies and focus groups as well as new recruits. Subjects will be given the device for home use for up to 60 days. Prior to entering the study all subjects will be screened for inclusion/exclusion criteria (Attachment 1). If subjects are eligible and wish to enter the study, they will complete an intake form (Attachment 2).

Subjects will be mailed the devices, adhesive rings (three different types), charger and instructional materials including Owner's Manual with appropriate indications, warnings and cautions, and Quick Start Guide to unbox at home. The attachment rings contain adhesives that are commercially available, are biocompatible, and approved for human use. Questions related to the unboxing are listed in attachment 3.

Once entered into the study users will be free to use the Soovu device as needed, with a recommendation to use daily. The phone app that controls the device automatically tracks the use of the device. Specifically, location of pain, which treatment profile (1-3) the subject used, relief post use, the time and number of uses per day, duration of each treatment, and whether the user viewed any of the supportive instructions contained on the app.

Subjects will periodically be contacted via telephone or internet and asked a set of questions and opinions . At the conclusion of the study subjects will be contacted via telephone or internet and asked a set of exit questions as well as to return the study device.

In addition, a social media site with participation limited to study participants will be made available for participants to share comments amongst themselves, and for the company to provide clarifications on product usage as needed.

Criteria for Evaluation of Safety Any adverse event related or unrelated to the tested products will be documented and reported as required (occurrence date, site, outcome and assessment of causality and severity etc.) following approved operating procedures. All adverse events will be recorded in the final study report. Adverse event instructions will be included in the participant's Informed Consent Statement and in the study materials.

Statistical Methods Data will be analyzed using analysis of variance with pain site, past treatments, and gender as discrete factors, and age as a covariate. Purchase interested will be assessed using frequency analysis.

ELIGIBILITY:
Inclusion Criteria:

* ● A total of 40 males and females aged 21-70, with recurring lower back will be recruited. Back pain sufferers must report pain at least 3 days/week for the past month. This back pain must be present for at least 6 months. Otherwise, self-reporting moderate good to excellent health;

  * Self-assessed pain intensity level 5 or greater on the 0-10 Numeric Pain scale. This corresponds to a mild to moderate pain intensity;
  * Having signed an Informed Consent Form (ICF), be able to read, comprehend, and sign the informed consent form;
  * Has Apple iPhone version 6 or later IOS operating system and willing to download device app
  * Available for the entire study duration;
  * Willing to comply with all study related requirements;

Exclusion Criteria:

* ● Has or had a history of clinically significant, severe, progressive, or uncontrolled renal, hepatic, hematological, immunologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, cerebrovascular or psychiatric disease;

  * Has sciatica where the sciatic component of the pain is greater than the non-radiating pain located in the low back;
  * Skin diseases and disorders (e.g., psoriasis, eczema, scars, wounds and other dermatological lesions…), which may prevent the location of the device to the skin;
  * Taking dietary supplements or herbal remedies inconsistently (on and off) for the month prior to enrollment. If taking these supplements, subjects must stay on a regular daily dose of the product(s) for the duration of the study. If not currently taking these supplements, subjects cannot start taking them during their participation in the study;
  * Patients with neoplasms receiving treatment that may interfere with the study;
  * Subjects who are self-reported to be pregnant, lactating or planning to become pregnant;
  * Having a history of hypersensitivity to similar products;

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06-15 (Estimated); Primary Completion 2020-09-20 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
pain level via numeric pain scale | After week 8 of treatment
  11 point Numeric pain scale

SECONDARY OUTCOMES:
Mood levels | After week 8 of treatment
  0-10 scale from Brief Pain Inventory
stress level | After week 8 of treatment
  0-10 scale from Brief Pain Inventory
Enjoyment of life | After week 8 of treatment
  0-10 scale BPI short form
Use of device | After week 8 of treatment
  Number of times per week device is used (0-70)
ease of use | After week 8 of treatment
  0-10 use scale
benefits scale | After week 8 of treatment
  0-10 scale from the Westendorp subscale
activity level | After week 8 of treatment
  0-10 scale from short form Brief Pain Inventory

CONTACTS AND LOCATIONS:
Overall Officials: charles chabal, MD, Principal Investigator — Soovu Labs

IPD SHARING:
Plan to Share IPD: No